CLINICAL TRIAL: NCT00736983
Title: Adalimumab for the Treatment of Perianal Fistulas in Crohn's Disease More Effective Alone or Combined to Ciprofloxacin
Brief Title: Adalimumab in Combination With Ciprofloxacin/Placebo Treatment of Perianal Fistulas in Crohn's
Acronym: Adafi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBD 08-01; EudraCT#: 2007-005832-10
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Crohn's Disease With Perianal Fistulas
Keywords: Perianal fistulas; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Adalimumab
  Interventions: Drug: adalimumab
- 2 (Placebo Comparator): ciprofloxacin
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: adalimumab — 24 weeks: 160 mg, 80 mg, and than 40mg every 2 weeks
  Other Names: Humira
  Arms: 1
Drug: ciprofloxacin — 12 weeks; daily 2 x 500mg
  Other Names: Cipro
  Arms: 2

SUMMARY:
To assess whether a combination of ciprofloxacin and adalimumab is more effective than adalimumab alone for the treatment of perianal fistulas in Crohn's disease

DETAILED DESCRIPTION:
Dutch multicenter, randomized, double-blind study with two arms. 146 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* proven Crohn's disease
* Single or multiple draining perianal fistulas

Exclusion Criteria:

* Abscesses
* Infliximab, cyclosporine, tacrolimus and antibiotics for Crohn's disease within past 3 months
* active viral infection
* significate cardiovascular dysfunction
* Pregnancy, Lactation
* Surgical bowel resection to be expected within 6 months
* Positive stool culture for enteric pathogens
* Total parental nutrition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Reduction of 50% or more from baseline to week 12 in the number of draining perianal fistulas. | 12 week

SECONDARY OUTCOMES:
Proportion of patients in remission | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: C.J. van der Woude, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (13):
- Netherlands (13):
  - AMC, Amsterdam
  - VU, Amsterdam
  - Deventer ziekenhuis, Deventer
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - UMC Gronigen, Groningen
  - LUMC, Leiden
  - AZ Maastricht, Maastricht
  - St Antonius ziekenhuis, Nieuwegein
  - UMC Radboud, Nijmegen
  - Erasmus MC, Rotterdam
  - Haga ziekenhuis, The Hague
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Dewint P, Hansen BE, Verhey E, Oldenburg B, Hommes DW, Pierik M, Ponsioen CI, van Dullemen HM, Russel M, van Bodegraven AA, van der Woude CJ. Adalimumab combined with ciprofloxacin is superior to adalimumab monotherapy in perianal fistula closure in Crohn's disease: a randomised, double-blind, placebo controlled trial (ADAFI). Gut. 2014 Feb;63(2):292-9. doi: 10.1136/gutjnl-2013-304488. Epub 2013 Mar 23. PMID 23525574